CLINICAL TRIAL: NCT06029621
Title: Comparison of Short-term and Longterm Outcomes Between Robot-assisted Thoracoscopy and Television-assisted Thoracoscopy Surgery Forthymoma : a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Robot-assisted vs VATS for Thymoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Deping Zhao, Administrative Director of Thoracic Surgery Department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STAR006
Record Dates: First submitted 2023-08-28; First posted 2023-09-08 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Thymoma
MeSH Terms: conditions — Thymoma | interventions — Thymectomy; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Intervention Model Description: RATS versus VATS
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RATS for Thymectomy (Experimental): The operator of the surgical incision and the route of entry were determined, and the endoscope and surgical instruments were inserted through the operating hole. The phrenic nerve and diaphragm began to gradually separate upward while avoiding nerve damage. Subsequently, the innominate vein was dissected to observe the branches of the thymus vessels and clamped with a 5 mm Hem-o-Lok clamp. Continue to dissect the left side of the thymus until near the phrenic nerve. After the thymus was removed entirely, it was placed in a bag and removed through an incision. After the operation, a 28 Fr chest tube was placed through the incision to the chest top. An 18 G central venous catheter was placed at the level of the posterior axillary line to the posterior costophrenic angle, and about 10 cm was inserted.
  Interventions: Procedure: RATS for Thymectomy
- VATS for Thymectomy (Active Comparator): The main operation principles and procedures of the operation are basically similar to those of the RATS and are completed under video-assisted thoracoscopic surgery.
  Interventions: Procedure: VATS for Thymectomy

INTERVENTIONS:
Procedure: RATS for Thymectomy — a minimally invasive surgical type for Thymoma: RATS
  Arms: RATS for Thymectomy
Procedure: VATS for Thymectomy — a minimally invasive surgical type for Thymoma: VATS
  Arms: VATS for Thymectomy

SUMMARY:
The aim of this study is to explore the advantages of robot-assisted thymectomy in long-term survival benefits and short-term clinical efficacy compared with video-assisted thoracoscopic thymectomy based on a multi-center, prospective, randomized controlled clinical trial.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery ( VATS ) is widely used in thoracic surgery and has gradually replaced traditional thoracotomy in thymoma. As a new type of VATS, the long-term oncological results of robot-assisted thoracoscopic surgery in thymoma have not been verified. Therefore, we designed a multicenter, prospective, randomized controlled clinical trial to determine whether RATS thymectomy is as effective as VATS thymectomy in terms of short-term and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. ) The age of the subjects on the day of signing the informed consent was ≥ 18 years old and < 75 years old, regardless of gender ;
2. ) Chest thin-layer CT and MR showed anterior mediastinal space-occupying lesions, combined with relevant hematological indicators, the patient was clinically diagnosed as a thymic epithelial tumor with or without myasthenia gravis ( MG ) symptoms.
3. ) need to accept thymectomy surgery ;
4. ) Clinical stage I to IIIA ( AJCC-UICC TNM staging system ) ;
5. ) The maximum diameter of the lesion < 5cm ;
6. ) physical condition score 0 or 1 ( Eastern Cooperative Oncology Group ECOG scoring system ) ;
7. ) Have not received any anti-thymoma therapy before, including but not limited to systemic chemotherapy, radiotherapy, etc. ;
8. ) Preoperative major organ function meets the following criteria : Bone marrow function: hemoglobin ≥ 10.0 g / dL ( no blood transfusion within 28 days before hemoglobin examination ), absolute neutrophil count ≥ 1.5 × 109 / L, platelet count ≥ 100 × 109 / L ( no transfusion of apheresis platelets or IL-11 treatment within 14 days before platelet count examination ) ; coagulation function : INR and PT < 1.5 × ULN, APTT ≤ 1.5 × ULN ; liver function: transaminase ( ALT and AST ) ≤ 2.5 × ULN; total bilirubin ≤ 1.5 × ULN ( Gilbert's syndrome or liver metastasis subjects total bilirubin ≤ 2.5 × ULN ) ; renal function: serum creatinine clearance rate ≥ 60 mL/min ( calculated according to the Cockcroft-Gault formula ) ;
9. ) voluntarily participated in and were able to undergo robot-assisted or thoracoscopic thymectomy, and complied with the study follow-up plan.

Exclusion Criteria:

1. ) Patients with myasthenia gravis crisis ;
2. ) had undergone mediastinal surgery or cardiac surgery ;
3. ) body mass index ( BMI ) ≥ 30 ;
4. ) Patients with severe liver and kidney dysfunction ( ALT and/or AST more than three times the upper limit of normal, Cr more than the upper limit of normal ) ;
5. ) combined with severe chronic lung diseases such as COPD, asthma, or interstitial lung disease ;
6. ) suffering from uncontrolled heart, kidney, gastrointestinal, and infectious diseases and other complications ;
7. ) patients with other malignant tumors or hematological diseases ;
8. ) combined with chronic pain or preoperative use of opioid analgesics ;
9. ) patients with thoracic deformity or combined with pectus carinatum and pectus excavatum ;
10. ) have mental disorders, such as anxiety disorders ;
11. ) pregnant and/or lactating women ;
12. ) is currently participating in other interventional clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2030-09-19 (Estimated); Study Completion 2030-09-19 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival (OS) | 5 year after surgery
  OS at 5 year after surgery

SECONDARY OUTCOMES:
Pain score | at 1 year after surgery
  Pain was assessed using a pain scale on the first day, 1 month, 6 months and 1 year after surgery. Pain was evaluated using the visual analogue scale (VAS) and the numerical rating scale (NRS), with higher scores indicating greater pain
quality of life (QOL) at 1 year by EORTC QLQ-C30 | at 1 year after surgery
  Quality of life was assessed at 1 month, 6 months and 1 year after surgery. QQL was evaluated using the European Organization for the Treatment and Research of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) version 3.0
quality of life (QOL) at 1 year by EQ-5D | at 1 year after surgery
  Quality of life was assessed at 1 month, 6 months and 1 year after surgery. QQL was evaluated using the European Five Dimensional Health Scale (EQ-5D).
R0 rate | postoperative in-hospital stay up to 30 days
  R0 radical rate
operative time | Intraoperative
  the time of operation
blood loss | Intraoperative
  blood loss in the operation
conversion rate | Intraoperative
  the rate of conversion to open surgery in the operation
length of hospital stay (LOS) | postoperative in-hospital stay up to 30 days
  length of stay in hospitalization
Catheterization days | postoperative in-hospital stay up to 30 days
  The interval days from the completion of catheter insertion to the removal of the thoracic tube
Volume of drainage | postoperative in-hospital stay up to 30 days
  Volume of drainage from the completion of catheter insertion to the removal of the thoracic tube
postoperative complications | postoperative in-hospital stay up to 30 days
  mainly include: pneumonia, arrhythmia, incision infection, vocal cord paralysis, trachea cannula
30-day mortality | postoperative in-hospital stay up to 30 days
  30-day mortality after surgery
30-day readmission rate after surgery | postoperative in-hospital stay up to 30 days
  Rate of readmission due to postoperative complications
5-year disease-free survival (DFS) | 5 year after surgery
  DFS at 5 year after surgery
Tumor recurrence rate | 5 year after surgery
  The rate of recurrence of thymoma in patients after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Deping Zhao, MD,PhD, Principal Investigator — Shanghai Pulmonary Hospital, School of Medicine, Tongji University
Locations (2):
- China (2):
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Zhejiang

IPD SHARING:
Plan to Share IPD: No